CLINICAL TRIAL: NCT04366180
Title: Multicentric Study to Assess the Effect of Consumption of Lactobacillus Coryniformis K8 on Healthcare Personnel Exposed to COVID-19
Brief Title: Evaluation of the Probiotic Lactobacillus Coryniformis K8 on COVID-19 Prevention in Healthcare Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P054
Record Dates: First submitted 2020-04-27; First posted 2020-04-28 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: Covid-19; Prevention; Healthcare workers
MeSH Terms: conditions — COVID-19 | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Experimental group who will receive one capsule of Lactobacillus K8 per day (3x10^9 cfu/day).
  Interventions: Dietary Supplement: Probiotic
- Control (Placebo Comparator): Control group who will receive a daily placebo capsule consisting of maltodextrin
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic group will received one capsule with Lactobacillus K8 per day (3x10^9 cfu/day) during 2 months
  Arms: Probiotic
Dietary Supplement: Control — The control group will received one placebo capsule per day during 2 months
  Arms: Control

SUMMARY:
The aim of the present study is to evaluate the effects of Lactobacillus coryniformis K8 consumption on the incidence and severity of Covid-19 in health workers exposed to the virus. This is a preventive study

ELIGIBILITY:
Inclusion Criteria:

1. Persons over 20 years of age.
2. Active healthcare personnel, who attend patients with COVID-19 disease, including all professional categories, medicine, nursing and warders.
3. Ability to complete surveys.
4. Signature of informed consent

Exclusion Criteria:

1. Person with positive test of COVID-19 confirmed by PCR test or serology
2. Person with concomitant pathology HIV, transplant, active oncology or other type of active immunosuppression
3. Pregnant women or women with intention to become pregnant in the next 2 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of SARS CoV-2 infection in healthcare workers | 8 weeks
  The incidence of SARS CoV-2 infection will be confirmed by PCR or antigen test

SECONDARY OUTCOMES:
Incidence of hospital admissions caused by SARS-CoV-2 infection | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), it will be evaluated how many of them will required hospital admission because of Covid-19
Incidence of ICU admissions caused by SARS-CoV-2 infection | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), it will be evaluated how many of them will required ICU admission because of Covid-19
Incidence of pneumonia caused by SARS-CoV-2 infection | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), it will be evaluated how many of them will develop pneumonia because of Covid-19
Incidence of oxygen support requirement caused by SARS-CoV-2 infection | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), it will be evaluated how many of them will require oxygen support because of Covid-19
Incidence of gastrointestinal symptoms caused by SARS-CoV-2 infection | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), it will be evaluated how many of them will develop gastrointestinal symptoms because of Covid-19
Days with body's temperature > 37.5 ºC | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), number of days with body's temperature > 37.5 ºC during the course of the disease
Days with cough | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), number of days with cough during the course of the disease
Days with fatigue | 8 weeks
  In the healthcare workers that confirm the SARS Cov-2 infection (primary variable), number of days with fatigue during the course of the disease
Medical treatment | 8 weeks
  Use of drugs (dosis and duration of the treatment) for Covid-19 treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Rodriguez Blanque, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Blanque R, Sanchez-Garcia JC, Cobos Vargas A, Leyva Martinez MS, Martinez Diz S, Cortes-Martin J, Tovar-Galvez MI. Evaluation of Lactobacillus Coryniformis K8 Consumption by Health Care Workers Exposed to COVID-19 (LactoCor2 Project): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 28;12:e37857. doi: 10.2196/37857. PMID 37285326